CLINICAL TRIAL: NCT00226460
Title: Phase 2, Double-blind, Randomized, Controlled Multi-center Clinical Trial of the Safety and Efficacy of Transplanted Fetal Porcine Cells in Patients With Parkinson's Disease.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Diacrin/Genzyme Corporation LLC (Industry)
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PD96-1101
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Drug: Fetal porcine cells, Neurocell-PD

SUMMARY:
The purpose of this study was to evaluate the differences in safety and efficacy between Parkinson's disease patients who either received transplantation of fetal porcine cells or placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient has idiopathic Parkinson's disease. a) with bradykinesia and either rest tremor or rigidity, b) history of asymmetry of Parkinson's disease signs, c) history of progression of Parkinson's disease signs, d) no other suspected cause of Parkinson's disease, e) the patient is L-DOPA responsive (based on the Treating Investigator's clinical judgment, the patient demonstrates a predictable ON response after the first daily dose of L-DOPA)
* The patient has had Parkinson's disease for at least 5 years (from onset of symptoms).
* The patient demonstrates unequivocal Clinical Off periods.
* Patient has been on a stable regimen of L-DOPA and any other anti-Parkinsonian medications for at least one month prior to start of screening.
* The patient demonstrates L-DOPA-or dopamine agonist-induced dyskinesias.
* The patient's age is 40-70.
* The patient is currently under "optimal medical therapy", as determined by the Treating Investigator.
* The patient has had a UPDRS assessment as per a modified CAPIT protocol at screening and the total UPDRS score in the defined OFF state was at least 60.
* If the patient is a woman of child bearing potential, she must not be nursing and an adequate form of birth control must be used for the duration of this trial.
* The patient has a normal chest x-ray and does not exhibit any signs or symptoms of coronary artery disease (on exam or on EKG) dysrhythmia (in order for surgery to be safely performed).
* The patient is able to understand and is willing to comply with study requirements; this may include travel within or outside the United States for neuroimaging testing and surgery. It will be necessary for a companion to travel with the patient.
* The patient is able to provide written informed consent.
* The patient understands that the Sponsor recommends that all patients in this trial avoid pregnancy and minimize the sharing of secretions with sexual partners.
* The patient is willing to participate in the life-long xenotransplantation registry.

Exclusion Criteria:

* The patient has a likely alternative diagnosis for Parkinsonism based on history, physical examination or laboratory testing. Atypical Parkinsonian variants (such as Shy-Drager, olivopontocerebellar atrophy, progressive supranuclear palsy and striatonigral degeneration) and secondary Parkinsonism (e.g., secondary to trauma or metabolic abnormalities; history of encephalitis, oculogyric crises or use of dopaminergic antagonists/depleting drugs) will be excluded.
* The patient has had a prior cranial neurosurgical procedure.
* The patient has MRI or CT evidence of abnormalities which could lead to Parkinsonism or make the patient an unsuitable neurosurgical candidate.
* The patient has a history of intracranial pathology (e.g., tumor, vascular malformation) that might make the patient an unsuitable neurosurgical candidate.
* The patient has a pre-existing medical condition that may interfere with the evaluation of the safety and/or effectiveness of the study agent or prevent study completion (e.g.:, symptomatic cardiac disease, impaired renal function or seizure disorder).
* The patient has a known sensitivity to products of porcine origin (e.g. pork).
* The patient has a known steroid or cyclosporine intolerance.
* The patient has significant cognitive impairment; specifically, a MMSE score of < 25, and, in the investigators judgment, the patient is demented.
* The patient has a Hamilton Depression score of > 16.
* The patient has hallucinations, delusions, psychosis or chronic psychiatric illness, with the exception of mild, L-DOPA induced hallucinations, or those caused by concomitant medications, which resolve with dose adjustment.
* The patient has a positive response to a tuberculin skin test (with the exception of patients who have either been inoculated for TB, or treated for the disease in the past).
* The patient has been treated during the 6 months prior to Screening with dopaminergic antagonists.
* (Females only) The patient is nursing or pregnant.
* The patient has taken tolcapone within 6 weeks of the Screening UPDRS exam.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-08; Study Completion 2001-01

PRIMARY OUTCOMES:
change in UPDRS

SECONDARY OUTCOMES:
change in PET scan

CONTACTS AND LOCATIONS:
Locations (1):
- PD and Movement Disorders, University of South Florida, Tampa, Florida, United States